CLINICAL TRIAL: NCT03178253
Title: Hypothyroidism in Patients With Type 2 Diabetes With Early Diabetic Nephropathy
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, maria hamdy, Assiut University, Assiut University
Other Study IDs: assuit1991
Record Dates: First submitted 2017-06-03; First posted 2017-06-06 (Actual); Last update posted 2017-06-07 (Actual); Status verified 2017-06

CONDITIONS: Hypothyroidism in Diabetes

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- 3

SUMMARY:
Diabetes Mellitus is the most common disorder seen. The impact of this disease on the quality of life, and on morbidity and mortality through the complications that affect the small and large vessels resulting in retinopathy, nephropathy, neuropathy, and ischemic heart disease has been emphasized by the findings of the national commission (USA) on diabetes .

So, there was curiosity to understand and learn the association of this disorder with another common endocrine gland function that is thyroid gland . The association between these two disorders has long been recognized although the prevalence of thyroid dysfunction in diabetic population varies widely between studies. With insulin and thyroid hormone being intimately involved in cellular metabolism and thus excess or deficit of these hormones result in functional derangement of the other.

DETAILED DESCRIPTION:
Diabetic patients have higher prevalence of thyroid disorder when compared with the normal population. Diabetic women are more frequently affected than men and hypothyroidism is more common than thyrotoxicosis .

Sub-clinical hypothyroidism is an independent risk factor for development of diabetic nephropathy. Severe hypothyroidism (biochemically) may be completely asymptomatic. Though our patient had throid stimulating hormone level more than 100 mIU/L, he did not have any symptoms of hypothyroidism.so diagnosis of hypothyroidism depends on laboratory parameters rather than clinical findings Recognition and treatment of hypothyroidism in diabetic patients will benefit glycemic control and improve general well-being ). Diabetic nephropathy, a major micro-vascular complication of type 2 diabetes mellitus, is an important cause of chronic kidney disease. It results from interactions between hemodynamic and metabolic factors .

ELIGIBILITY:
Inclusion Criteria:

* All patients with Type 2 diabetes mellitus and with diabetic nephropathy.
* All diabetics irrespective of glucose control.
* All diabetics irrespective of treatment (oral hypoglycemic drugs/insulin)

Exclusion Criteria:

* 1) Type 1 diabetes mellitus 2) Patients with:

  * Gestational diabetes mellitus.
  * Pancreatitis.
  * Steroid induced Diabetes.
  * hepatobiliary disease
  * on systemic drug therapy such glucocorticoids and oral contraceptives.

Ages: 40 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: all diabetic patients
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2017-06-30 (Estimated); Primary Completion 2017-06-30 (Estimated); Study Completion 2018-06-30 (Estimated)

PRIMARY OUTCOMES:
percentage of hypothyroidism in patients of type 2 diabetes with diabetic nephropathy | one year

CONTACTS AND LOCATIONS:
Locations (1):
- Maria Hamdy, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided